CLINICAL TRIAL: NCT07322094
Title: CATALINA-4: Phase 1B/2 Study of TORL-1-23 With Neoadjuvant Chemotherapy and Interval Cytoreductive Surgery in Newly Diagnosed Patients With Advanced Stage Ovarian Cancer
Brief Title: CATALINA-4: A Study to Investigate the Safety and Efficacy of TORL-1-23 With Chemotherapy Given Before Initial Surgery in Women With Advanced Stage Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TORL Biotherapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TORL123-004
Record Dates: First submitted 2025-12-17; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: FIGO Stage III and IV Ovarian Cancer; Fallopian Tube Cancers; Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm A: TORL-1-23 and paclitaxel (Experimental): Administered once every three weeks
  Interventions: Combination Product: TORL-1-23 and paclitaxel
- Treatment Arm B: TORL-1-23 and carboplatin (Experimental): Administered once every three weeks
  Interventions: Combination Product: TORL-1-23 and carboplatin
- Treatment Arm C: TORL-1-23, paclitaxel, and carboplatin (Experimental): Administered once every three weeks
  Interventions: Combination Product: TORL-1-23, paclitaxel, and carboplatin

INTERVENTIONS:
Combination Product: TORL-1-23 and paclitaxel — TORL-1-23 and paclitaxel
  Arms: Treatment Arm A: TORL-1-23 and paclitaxel
Combination Product: TORL-1-23 and carboplatin — TORL-1-23 and carboplatin
  Arms: Treatment Arm B: TORL-1-23 and carboplatin
Combination Product: TORL-1-23, paclitaxel, and carboplatin — TORL-1-23, paclitaxel, and carboplatin
  Arms: Treatment Arm C: TORL-1-23, paclitaxel, and carboplatin

SUMMARY:
A Phase 1B/2 Study to Investigate the Safety and Efficacy of TORL-1-23 with Chemotherapy Given Before Initial Surgery in Women with Advanced Stage Ovarian Cancer

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Histologically or cytologically confirmed diagnosis of epithelial ovarian, primary peritoneal or fallopian tubes cancer
* FIGO Stage III or IV
* Positive for claudin 6 (CLDN6) expression
* Adequate organ function

Exclusion Criteria:

* Clear cell, mucinous, sarcomatous, mixed histology, low-grade/borderline, or non-epithelial ovarian cancers
* Prior systemic treatment for the disease under study
* Prior surgery
* Prior radiation therapy to the abdomen or pelvis
* Current recipient or receipt within 5-half-lives of C1D1 of chemotherapy, biologic/targeted therapy, immunomodulator therapy for any disease indication
* Active, progressive, or symptomatic brain metastases
* Participants considered poor medical risks due to serious, uncontrolled medical conditions, active infections, or nonmalignant systemic diseases
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety and feasibility of TORL-1-23 in combination with chemotherapy by analyzing the incidence of treatment emergent adverse events and serious adverse events. | Treatment during Cycle 1 to Cycle 4 (Each cycle is 21 days)
  Incidence of Grade greater than or equal to 3 (using CTCAE V5.0) treatment-emergent adverse event (TEAE) and related serious adverse event (SAE)
To assess the efficacy of neoadjuvant TORL-1-23 in combination with chemotherapy | postoperative after Cycle 4 (Each cycle is 21 days)
  Determination of percentage CRS3 score for each treatment arm

SECONDARY OUTCOMES:
To assess the tolerability of TORL-1-23 in combination with chemotherapy | Treatment up to Cycle 8 (each cycle is 21 days)
  Safety assessed by incidence of intolerable Grade 2 and Grade greater than or equal to 3 TEAE and related SAE.
To characterize duration of benefit for TORL-1-23 plus chemotherapy | Measured up to 15 months after surgery
  Relapse free survival for participants

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No